CLINICAL TRIAL: NCT00547235
Title: Protocol For The Emergency Use Of Adoptive Immunotherapy With CMV-Specific T Cells Following HLA-Matched Unrelated Donor Bone Marrow Transplant Of An Infant With ADA-SCIDs And Pre Transplant CMV Infection
Brief Title: Emergency Use of Adoptive Immunotherapy With CMV-Specific T Cells After Donor Bone Marrow Transplant of an Infant With Immunodeficiency Syndrome and CMV Infection
Status: No longer available | Type: Expanded Access
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Thomas Manley, MD, Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Other Study IDs: 2215.00; FHCRC-2215.00; CDR0000570998 (Registry Identifier: PDQ)
Record Dates: First submitted 2007-10-19; First posted 2007-10-22 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2010-08

CONDITIONS: Infection; Precancerous/Nonmalignant Condition
Keywords: infection; precancerous/nonmalignant condition
MeSH Terms: conditions — Infections; Precancerous Conditions | interventions — Whole-Body Irradiation

INTERVENTIONS:
Biological: therapeutic allogeneic lymphocytes
Procedure: allogeneic bone marrow transplantation
Radiation: total-body irradiation

SUMMARY:
RATIONALE: Collecting the T cells from a donor and transplanting them into a patient may be effective treatment for immunodeficiency syndrome and CMV infection.

PURPOSE: This clinical trial is studying the emergency use of adoptive immunotherapy with CMV-specific T cells after donor bone marrow transplant of an infant with immunodeficiency syndrome and CMV infection.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine if adoptive immunotherapy with donor-derived CD4+ and CD8+ CMV- specific cytotoxic lymphocyte cell lines can augment T-cell immunity and treat CMV infection post transplant in a patient with severe combined immunodeficiency syndrome.

OUTLINE: The patient will undergo HLA-matched unrelated donor bone marrow transplantation from a CMV-seropositive donor after undergoing conditioning with 200cGy total-body irradiation per protocol FHCRC Protocol 1227.

CD8-positive and CD4-positive CMV-specific T cells are collected from the donor and used to generate T-cell lines.

If the patient has progressive or persistent CMV infection, then she will receive donor T cells IV over 30 minutes. Infusions may be repeated after at least 14 days if the previous infusion was well tolerated and if the CMV infection is persistent or increasing.

The patient undergoes blood sample collection at baseline and 7 days after T-cell infusion to assess CMV-specific T-cell response.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Adenosine deaminase-deficient severe combined immunodeficiency syndrome (ADA-SCIDs)
* CMV interstitial pneumonia based on the constellation of clinical and radiological findings

PATIENT CHARACTERISTICS:

* Female
* Oxygen desaturation (pulse oximetry 85% on room air)
* Abnormal chest radiograph
* No CMV retinitis

PRIOR CONCURRENT THERAPY:

* Prior ganciclovir and foscarnet sodium

Max Age: 1 Year | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2007-09; Primary Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Manley, MD, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States